CLINICAL TRIAL: NCT01638689
Title: A PET Study to Determine Alterations in Serotonin Levels in Human Brain After a Single Dose of Escitalopram
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magdalena Nord, MD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-019363-11; 2010-019363-11 (EudraCT Number)
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Mechanism of Action of escitalopram
MeSH Terms: interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 20 mg p.o.

SUMMARY:
Healthy males were examined with positron emission tomography (PET) and the radioligand 11C-AZ10419369, before and after administration of a single dose escitalopram. A change in the binding potential of 11C-AZ10419369 between the baseline and the post-dose condition was hypothesized to reflect a change in serotonin concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male gender
3. Age 20 to 30 years
4. Healthy according to physical examination, ECG, MRI and blood chemistry

Exclusion Criteria:

1. Past or present psychiatric disease
2. Past or present brain disorder or injury, including loss of consciousness for more than five minutes
3. Past or present drug or alcohol abuse
4. Past or present use of antidepressant or antipsychotic medications
5. Regular use of medications (including herbals), that could interfere with the pharmacodynamics or pharmacokinetics of escitalopram
6. Significant abnormality on ECG
7. Structural abnormality in the brain confirmed by MR examination
8. Claustrophobia
9. Any metal devises or implants in the body
10. Intolerance to escitalopram or any of the components of the formula
11. Predisposition to motion sickness
12. Inability to understand and comply with the study requirements
13. Any medical condition that, in the opinion of the investigator, make the subject unsuitable for the study or put the subject at additional risk

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in binding potential of 11C-AZ10419369 between baseline and post-dose condition | One day (PET measurement before and after escitalopram administration on the same day)

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Nord, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- PET center, Department of Clinical neuroscience, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Nord M, Finnema SJ, Halldin C, Farde L. Effect of a single dose of escitalopram on serotonin concentration in the non-human and human primate brain. Int J Neuropsychopharmacol. 2013 Aug;16(7):1577-86. doi: 10.1017/S1461145712001617. Epub 2013 Jan 25. PMID 23351590